CLINICAL TRIAL: NCT03089021
Title: Maitland Mobilization Versus Mulligan Mobilization in Sub-Acute and Chronic Non-Specific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Samar Mohammed Alansari, physical therapist, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB -PGS-2016-03-143
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Nonspecific Neck Pain
Keywords: neck pain,
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mulligan mobilization (Experimental): mobilization for spinous process or facet with neck movement 10 repetetions for 3 times.
  Interventions: Other: mulligan mobilization
- maitland mobilization (Experimental): maitland mobilization for spinous process or facet joint for 2 min and repeated 3 times.
  Interventions: Other: maitland mobilization

INTERVENTIONS:
Other: mulligan mobilization — mobilization with movement for spinous process or facet joint.
  Arms: mulligan mobilization
Other: maitland mobilization — posterioanterior of spinous process or facet joint.
  Arms: maitland mobilization

SUMMARY:
This study investigate the short term effect of Maitland in comparison to Mulligan mobilization with sub-acute and chronic non specific neck pain to improve neck pain, pain pressure threshold, rang of motion, joint position sense, disability, and to evaluate the interaction with psychological factors.

Study design: experimental study

DETAILED DESCRIPTION:
44 patients with sub-acute or chronic neck pain will be randomized into Maitland group: 22 patients receive central postro anterior or unilateral postero anterior. Mulligan group: 22 patients receive sustain natural apophyseal glides. The treatment will be 2 times /week for three weeks. Measurement will be taken pre intervention and after three weeks for neck pain, pain pressure threshold, range of motion, joint position sense, and disability using a numeric pain rating scale, pain pressure threshold test, cervical range of motion device, and neck disability index, depression, anxiety, fear avoidance believe and pain catestrophizing respectively.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged between 20 to 50 years.

  * Neck pain more than one week without radicular symptoms.
  * Pain on posterior neck from superior nuchal line to first thoracic vertebra.

Exclusion Criteria:

* • Patient contraindicate to mobilization (pregnancy, whiplash injury, tumor, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis and resting blood pressure higher than 140/90 mmHg).

  * Cervical radiculopathy.
  * Fibromyalgia pain syndrome.
  * Previous neck surgery.
  * Neck pain associate with vertigo caused by vertebrobasilar insufficiency or chronic headache.
  * Patient received physical therapy treatment in the previous three months.
  * Psychiatric disorders.
  * Vestibular system deficits.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-12-28 (Estimated)

PRIMARY OUTCOMES:
pain pressure threshold | 3 weeks
  It will be measured with an electronic algometer (Somedic AB, Farsta, Sweden) with a circular probe of 1 cm2. The PPT will be measured over the following site: (1) area of maximum tenderness over the cervical spine as identify by palpation, (2) tibialis anterior muscle (upper one-third of the muscle belly) bilateral. Tibialis anterior sites will be as remote lower limb sites to investigate any widespread changes in sensitivity. The pressure will be applied perpendicular over the identified sites at a rate of 40 KPa/s until the individual verbally states that the pressure is starting to change to a pain sensation. Then, the pressure will be stopped. The test will be repeated three times for each site within 30 second between measurements. An average of three measurements will be calculated
pain intensity | 3 weeks
  : numeric pain rating scale (NPRS) will be used to evaluate the intensity of pain perceived by patient. Pain is rated on 11 point scale from (0) no pain to (10) sever pain. The patients will be asked to point out the number that describes their pain level.

SECONDARY OUTCOMES:
cervical range of motion | 3 weeks
  it will be measured by cervical range of motion (CROM) device. It consists of three gravitational inclinometers system for flexion, extension and lateral flexion, and magnetic inclinometer for rotation.
joint position sense | 3 weeks
  it will be measured by using the (CROM) device
neck disability index | 3 weeks
  This questioner is used to report disability results from neck pain and it is a self-report based outcome. In addition, it contains ten sections with total score of 50 points

OTHER OUTCOMES:
State trait anxiety inventory questionnaire (STAI-Y): | 3 weeks
  It has 20 items for assessing trait anxiety and 20 for state anxiety
Beck depression inventory questionnaire (BDI) | 3 weeks
  it contains 21 items; each item has four self evaluation statements in a time frame of two weeks, and scores from 0 to 3. The total score for 21 items range from 0 to 63
Fear avoidance believe questionnaire (FABQ) | 3 weeks
  this questionnaire can assess the fear avoidance believe about the pain. It consists of 16 items. First five questions are related to fear avoidance of physical activities (FABQ- PA). Then the eleven questions are related to avoidance of work (FABQ-W). The score for each question is ranged from 0 (strong disagreement) to 6 (strong agreement). The total score is ranged from 0 to 66. Higher score is represented high level of fear avoidance believe
pain catestrophizing scale | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: samar alansari, master, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Abdulaziz Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
only coded data (describtive)